CLINICAL TRIAL: NCT03564639
Title: Hepatitis C Reinfection in an Injection Drug Using Population in Kenya: A Follow-up to the TLC-IDU Hepatitis C V Supplement Study.
Brief Title: Examining Hepatitis C Reinfection Rates in Kenya
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1512016965_B
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Research staff will obtain a sample of capillary or venous blood from participants at the treatment site and send specimens to Kenya Medical Research Institute (KEMRI) laboratory in Kisumu, Kenya for a Hepatitis C V RNA test. If viral load is detectable confirmatory samples will be sent to the Center for Disease Control (CDC) laboratory for next generation sequencing, to guide treatment. Samples will be collected at two time points post SVR and if re-treated in this study, 12 weeks after treatment completion to determine SVR.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Injection drug users with HCV: People who inject drugs who were confirmed positive for HCV and initiated treatment in the parent study beginning in September 2017.

SUMMARY:
The goal of this research project is to build upon the Testing and Linkage to Care for Injecting Drug Users (TLC-IDU) parent study and describe post-cure HCV reinfection in a population of people who inject drugs (PWIDs) in Kenya.

DETAILED DESCRIPTION:
In addition to describing reinfection in a substance using cohort, we will identify individual predictors of HCV reinfection in Kenya, as well as identifying individual utilization intervention approaches and dosing that reduce reinfection risk and treatment cite level risk factors (frequency of visits, community vs hospital location etc.). Determining the risk factors specific to reinfection and understanding the impact of concurrent harm reduction interventions will guide service delivery and implementation of HCV elimination strategies in Kenya and throughout the region.

ELIGIBILITY:
Inclusion Criteria:

1. Live in Nairobi or coastal Mombasa (Coast Province including Malindi), Kenya;
2. Are injection drug users (IDUs) that ever injected any non-prescribed drugs; and able and willing to provide informed consent.
3. Participates are in the parent study;
4. Complete treatment protocol; and achieve a sustained virologic response (SVR).

Exclusion Criteria:

Not in the above inclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study is taking place in the Mombasa province in Coastal Kenya and Nairobi, Kenya's capital. Participants were also in the parent study, were infected with HVC, have completed HVC treatment.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
HCV Reinfection | 6-18 months post sustained virologic response (SVR) to HCV treatment.
  The reinfection of patients with hepatitis C after completion of a previous HCV infection treatment.
Evaluate psychoeducational counseling | 6 months
  Brief questionnaire on knowledge, attitude and beliefs of each participant.
Examine usage of methadone maintenance | 12 months
  Brief questionnaire on services used
Examine usage of needle exchange programs | 12 months
  Brief questionnaire on services used
Evaluate psychoeducational counseling | 12 months
  Brief questionnaire on knowledge, attitude and beliefs of each participant.

SECONDARY OUTCOMES:
HCV reinfection referrals for treatment at Kenyetta National Hospital | 9-16 months post treatment
  Confirmed HCV reinfection cases will receive referrals to Kenyatta National Hospital and Coast General Hospital for treatment and management.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Kurth, PhD, Principal Investigator — Yale University School of Nursing
Locations (1):
- NASCOP, Nairobi, Kenya